CLINICAL TRIAL: NCT05924477
Title: Glaucoma Drainage Device and Endothelial Cell Loss Compare Trial
Acronym: DECLARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Eye Institute (NEI) (NIH); University of California, San Francisco (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 853474; UG1EY033703 (NIH)
Record Dates: First submitted 2023-06-08; First posted 2023-06-29 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Glaucoma
Keywords: glaucoma; glaucoma drainage device; endothelial cell density; endothelial cell loss; intraocular pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: A prospective 1:1 randomized, parallel design, double-masked clinical trial. Stratification is by clinical center and type of surgery (GDD alone vs GDD combined with phacoemulsification).
Who Masked: Participant, Outcomes Assessor
Masking Description: All trial participants will be masked to their tube locations. The primary outcome accessors who grade specular microscopy images at the PRC, perform IOP measurements at each clinical center, or conduct the MDS analysis at the Metagenomic RNA Deep Sequencing (RNA-seq) Center will also be masked to tube locations. Due to the nature of the surgical intervention, the surgeon, the technician taking specular microscopy and AS-OCT images, and the graders at the PRC who will perform AS-OCT measurements will not be masked to the tube locations. However, the graders of AS-OCT images will be masked to the purpose of the study and will be different from the graders of specular microscopy images.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulcus tube placement (Active Comparator): Glaucoma drainage device (GDD) implantation with tube placement in the ciliary sulcus
  Interventions: Procedure: Sulcus tube placement
- Anterior chamber (AC) tube placement (Active Comparator): Glaucoma drainage device (GDD) implantation with tube placement in the anterior chamber
  Interventions: Procedure: Anterior chamber (AC) tube placement

INTERVENTIONS:
Procedure: Sulcus tube placement — GDD implantation surgery with tube placement in the ciliary sulcus
  Arms: Sulcus tube placement
Procedure: Anterior chamber (AC) tube placement — GDD implantation surgery with tube placement in the anterior chamber
  Arms: Anterior chamber (AC) tube placement

SUMMARY:
Glaucoma Drainage Device and Endothelial Cell Loss Compare Trial (DECLARE) is a multi-center, outcome-masked, randomized clinical trial. The purpose of this study is to compare glaucoma drainage device implantation in the anterior chamber (front part of the eye) and sulcus (small space between iris and front chamber of the eye) in efforts to minimize cell loss in the eye.

DETAILED DESCRIPTION:
The DECLARE Trial is a prospective 1:1 randomized, parallel design, double-masked clinical trial to compare endothelial cell density (ECD), intraocular pressure (IOP) and metagenomic RNA deep sequencing (MDS) between sulcus and anterior chamber (AC) tube placement after glaucoma drainage device (GDD) implantation.

The trial has fixed sample size with 12 months follow-up for primary outcome assessment and trial participants will continue to be followed to the end of grant cycle with a total of 24 months follow-up.

Patients will be randomized to 2 tube locations for GDD implantation:

* Tube placed in the AC
* Tube placed in ciliary sulcus
* Stratification: by clinical center and type of surgery (GDD alone vs GDD combined with phacoemulsification). Stratified randomization by clinical center is to ensure that a similar number of subjects will be randomized to either sulcus tube or AC tube placement for a specific clinical center. Because eyes undergoing a combined phacoemulsification with GDD implantation may be associate with larger ECL from phacoemulsification, stratified by surgery type is to ensure two tube location groups similar number of study eyes that will undergo a combined phacoemulsification with GDD implantation.

ELIGIBILITY:
Inclusion Criteria:

* Medically uncontrolled glaucoma requiring GDD or GDD combined with phacoemulsification as the planned surgical procedure
* Candidate for GDD implantation for ciliary sulcus and AC tube
* Age greater than or equal to 18 years old

Exclusion Criteria:

* Preexisting corneal condition that would affect the corneal endothelium or previous corneal transplant
* Presence or history of Cypass Micro-Stent
* Previous GDD, Xen Gel Stent or Preserflo MicroShunt removed less than 6 months before surgery
* Presence of GDD implantation, Xen Gel Stent, of Preserflo MicroShunt
* Previous trabeculectomy and/or minimally invasive glaucoma surgery within the past 6 months
* AC intraocular lens
* Presence of nanophthalmos, uncontrolled uveitis, silicone oil, Sturge-Weber syndrome or other conditions associated with elevated episcleral venous pressure
* Unwilling or unable to give consent, unwilling to accept randomization, or unable to return for scheduled protocol visits
* No light perception vision in the study eye or fellow eye visual acuity < 20/200
* Need for glaucoma surgery combined with other ocular procedures (i.e. corneal transplant, or retinal surgery) or anticipated need for additional ocular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Central endothelial cell loss (ECL) from baseline | Baseline to 12 months
  Change in central endothelial cell density based on assessment of Specular Microscopy images.

SECONDARY OUTCOMES:
Intraocular Pressure (IOP) at 12 months | 12 months after GDD implantation
  Goldman applanation tonometry (preferred method)
ECD at 12 months after GDD implantation | 12 months after GDD implantation
  ECD measures will be based on the assessment of Specular Microscopy images
Best-corrected visual acuity (BCVA) at 12 months after GDD implantation | 12 months after GDD implantation
  Distance BCVA using an ETDRS eye chart and recorded as number of letters read correctly.
Number of anti-glaucoma medications at 12 months after GDD implantation | 12 months after GDD implantation
  Topical and oral anti-glaucoma medication information is collected at all visits.

OTHER OUTCOMES:
MDS (Metagenomic RNA Deep Sequencing) analysis at 12 months | 12 months after GDD implantation
  Gene profile analysis evaluating anterior chamber microenvironment (by collecting aqueous fluid samples from the study eye)
Central endothelial cell loss (ECL) from baseline | Baseline to 24 months
  Change in central endothelial cell density based on assessment of Specular Microscopy images.
Intraocular Pressure (IOP) at 24 months | 24 months after GDD implantation
  Goldman applanation tonometry (preferred method)
ECD at 24 months after GDD implantation | 24 months after GDD implantation
  ECD measures will be based on the assessment of Specular Microscopy images
Best-corrected visual acuity (BCVA) at 24 months after GDD implantation | 24 months after GDD implantation
  Distance BCVA using an ETDRS eye chart and recorded as number of letters read correctly.
Number of anti-glaucoma medications at 24 months after GDD implantation | 24 months after GDD implantation
  Topical and oral anti-glaucoma medication information is collected at all visits.
Safety outcomes: surgical complications | At the GDD surgery visit, and up to 24 months after GDD implantation
  All AEs, including hypotony, hyphema, tub-related complications, tube exposure, choroidal detachment, corneal decompensation, endophthalmitis and others.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, MD, PhD, Study Chair — University of California, San Francisco; Jennifer Rose-Nussbaumer, MD, Study Director — Stanford University; Thuy Doan, MD, PhD, Study Director — University of California San Fransicso
Locations (8):
- United States (7):
  - University of California San Francisco, San Francisco, California
  - Diablo Eye Associates, Walnut Creek, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Wilmer Eye Institute, Johns Hopkins University, Baltimore, Maryland
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - University of Buffalo/State University of New York, Buffalo, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- Prism Eye Institute, University of Toronto, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No